CLINICAL TRIAL: NCT05709171
Title: Dual 64Cu-DOTATATE and 18F-FDG PET/CT Imaging of Patients With Neuroendocrine Neoplasms
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mathias Loft, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK_NEN_DOTA-FDG_21
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: GEP-NET; Neuroendocrine Tumors; Neuroendocrine Carcinoma; Neuroendocrine Carcinoma Metastatic
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — Fluorodeoxyglucose F18; 64Cu-DOTATATE; Copper; copper dotatate CU-64

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Each patient will undergo one standard of care 18FDG PET/CT and one 64Cu-DOTATATE PET/CT within 4 weeks.
  Interventions: Drug: 18F-FDG; Drug: 64Cu-Dotatate

INTERVENTIONS:
Drug: 18F-FDG — PET/CT scan approximately 60 min after injection of 18F-FDG
  Other Names: 18F-fluorodeoxyglucose; fluorodeoxyglucose-F-18; [18F]F-FDG
Drug: 64Cu-Dotatate — PET/CT scan approximately 60 min after injection of 64Cu-Dotatate
  Other Names: Copper (64Cu) oxodotreotide

SUMMARY:
Prospective clinical trial investigating combined, dual 18F-FDG PET/CT and 64Cu-DOTATATE PET/CT imaging of patients with gastroenteropancreatic neuroendocrine neoplasms (GEP-NEN)

DETAILED DESCRIPTION:
Patients with neuroendocrine neoplasms (NEN) represent a heterogeneous disease group with variable prognosis. NEN most frequently arise from the gastrointestinal tract or the pancreas; collectively termed GEP-NEN. Grading of GEP-NEN is based on tumor proliferation index (Ki-67) from biopsies or surgical resection specimens into: low grade G1 neuroendocrine tumor (NET) (Ki-67<3%), intermediate grade G2 NET (Ki-67 3-20%) and high grade NEN (Ki-67%>20). High grade NENs are further categorized according to tissue morphology into well-differentiated G3 neuroendocrine tumors (NET) and poorly differentiated neuroendocrine carcinomas (NEC).

A common feature of most NETs is the overexpression of somatostatin receptors (SSR) on the tumor cell surface. Whole-body PET/CT imaging with radiolabelled SSR-targeted tracers, e.g. 64Cu-DOTATATE, plays a key role in diagnosis, staging, treatment selection and response evaluation of patients with NET. Measurements of 64Cu-DOTATATE tumor standardized uptake values (SUV) and tumor volume on PET/CT provide prognostic value for patients with NET. Patients with high grade NEN often have lower SSR expression and SSR PET/CT is infrequently routinely performed in these patients. However, we expect that the SUV and tumor volume from 64Cu-DOTATATE PET/CT also holds prognostic information for patients with high grade NEN and that some patients may prove eligible for PRRT based on the scans.

18F-FDG PET/CT imaging is widely used in cancers, but is routinely primarily reserved for patients with high grade NEN. However, 18F-FDG PET/CT also holds prognostic information for patients with lower grade NET.

By combining 64Cu-DOTATATE PET/CT and 18F-FDG PET/CT imaging, we expect to obtain complementary prognostic information for patients with GEP-NEN of all grades. In this clinical trial, we will therefore investigate and compare the tumor phenotypes found on 64Cu-DOTATATE PET/CT and 18FDG PET/CT performed within 4 weeks in patients with GEP-NET G1-3 and GEP-NEC. The aim of the trial is to establish prognostic models for progression-free-survival (PSF) and overall survival (OS) including tumor status (positive/negative), SUV measurements, and tumor volume derived from the dual 64Cu-DOTATATE PET/CT and 18FDG PET/CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically verified gastro-entero-pancreatic neuroendocrine neoplasm (GEP-NEN) or patients with unknown primary tumor with metastases with verified NEN positive histopathological examination suggesting GEP origin
* World Health Organization (WHO) Performance status 0-2
* Must be able to read and understand the patient information in Danish and to give informed consent

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Weights more than the maximum weight limit for the PET/CT bed of the scanner (140 kg)
* Uncontrolled diabetes
* Uncontrolled infection
* Exacerbation in autoimmune diseases
* Other active cancer disease
* Conditions or diseases (e.g. uncontrolled Parkinson's disease) making the patient unable to lie still in the scanner
* Severe claustrophobia
* Localized neuroendocrine neoplasms of the appendix, the rectum measuring < 1 cm, and ECL-omas of the stomach
* History of allergic reaction attributable to compounds of similar chemical or biologic com-position to 18FDG or 64Cu-DOTATATE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 12 months after last-patients-last-visit
  Time to disease progression from PET/CT scans. Disease progression is defined as a composite measure (whichever occurs first) of RECIST-1.1 defined radiological progression, commencement of another systemic therapy and/or surgery/embolization/ablation related to worsening to the patient's disease status after the index scan, progression evaluated by a multidisciplinary tumor board, and death related to the patient's NEN disease. In case of uncertainty if progression has occurred, the patient's disease status will be evaluated by a multidisciplinary tumor board.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 months after last-patients-last-visit
  Time to death from PET/CT scans.
Correlation between tumor standardized uptake values (SUV) on 18F-FDG PET and 64Cu-DOTATATE PET | 12 months after last-patients-last-visit
  SUV measured on matched tumors on 18F-FDG PET and 64Cu-DOTATATE PET are compared
Proportion of patients eligible for peptide receptor radionuclide therapy (PRRT) | 12 months after last-patients-last-visit
  The proportion of patients who are considered eligible for PRRT based on their 64Cu-DOTATATE PET/CT according to the routine clinical guidelines at the department

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjaer, MD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not publicly available due to protection of personal data according to data protection regulations and medical confidentiality.